CLINICAL TRIAL: NCT04113668
Title: AN OPEN-LABEL, SINGLE-SEQUENCE, CROSSOVER STUDY TO INVESTIGATE THE EFFECTS OF UGT1A9 INHIBITOR DIFLUNISAL, AT STEADY-STATE, ON PHARMACOKINETICS OF A SINGLE DOSE OF BMS-986165 IN HEALTHY MALE AND FEMALE VOLUNTEERS
Brief Title: The Effects Diflunisal on the Levels of BMS-986165 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: IM011-101
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Healthy Participants
MeSH Terms: interventions — deucravacitinib; Diflunisal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Single Dose (BMS-986165) (Experimental)
  Interventions: Drug: BMS-986165
- Arm B:Diflunisal and Single Dose (BMS-986165) (Experimental)
  Interventions: Drug: BMS-986165; Drug: diflunisal

INTERVENTIONS:
Drug: BMS-986165 — Specified Dose on Specified Days
Drug: diflunisal — Specified Dose on Specified Days
  Arms: Arm B:Diflunisal and Single Dose (BMS-986165)

SUMMARY:
BMS-986165 Is broken down by the body through multiple pathways. This study Investigates the effect of blocking one pathway in the drug levels of BMS-986165 in health subjects.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Women and men must agree to follow instructions for methods of contraception.
* Participants must be willing and able to complete all study-specific procedures and visits.
* A healthy participant, as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations.
* WOCBP must have a negative serum or urine pregnancy test within 24 hours prior to the start of study treatment.

Exclusion Criteria:

* Any significant acute or chronic medical condition that presents a potential risk to the participant and/or may compromise the objectives of the study, including a history of active liver disease
* History of biliary disorders, including Gilbert's syndrome or Dubin- Johnson disease, in addition to, current or recent gastrointestinal disease that could impact the absorption of study drug.
* Participants using electronic cigarettes or nicotine-containing products who have stopped smoking less than 6 months prior to dosing on Day 1.
* Consumption of chargrilled meat, quinine, or any nutrient known to modulate CYP enzyme activity within 14 days prior to first administration of study treatment.
* History of any significant drug allergy

Other inclusion/exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986165 with and without UGT1A9 inhibitor | Up to 14 days
Area under the plasma concentration-time AUC (0-T) of BMS-986165 with and without UGT1A9 inhibitor | up to 14 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time AUC(INF) for BMS-986165 with and without UGT1A9 inhibitor | up to 14 days

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | up to 48 days
Number of participants with 12-lead Electrocardiogram (ECG) Abnormalities | up to 48 days
Physical Examination of weight | up to 48 days
Number of changes in blood pressure | up to 20 days
Number of changes in body temperature | up to 20 days
Number of changes in respiratory rate | up to 20 days
Number of clinical significant changes in lab assessment of blood serum | up to 48 days
Number of Clinically significant changes in assessment of blood | up to 20 days
Number of Clinically significant changes in lab assessment of urine | up to 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PRA Health Sciences - Lenexa, Lenexa, Kansas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm